CLINICAL TRIAL: NCT07397741
Title: Evaluation of CCR6 Gene Expression and Circulating CCL20 Levels as Potential Biomarkers in Rheumatoid Arthritis
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Salma Khalaf Abdelmageed, Assistant lecturer of medical biochemistry, Sohag University
Other Study IDs: Soh-Med-26-1-3MD
Record Dates: First submitted 2026-01-30; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Rhematoid Arthritis
Keywords: CCR6/CCL20 axis in Rheumatoid arthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: Patients with Rheumatoid Arthritis
  Interventions: Genetic: Gene expression by quantitative Real Time PCR
- Group II: apparently healthy controls with no chronic illness of matched age and sex
  Interventions: Genetic: Gene expression by quantitative Real Time PCR

INTERVENTIONS:
Genetic: Gene expression by quantitative Real Time PCR — Sample collection:
  * 5 ml peripheral blood will be collected under sterile conditions.
    1-Gene Expression Assay
  * Total RNA Extraction
  * cDNA Synthesis
  * Gene Expression Analysis:
    o Quantitative Real-Time PCR (qRT-PCR) for CCR6 gene expression using primer as follows: Forward primer (5'-3'): CCACAATGAGCGGGGAATCAATGAA Reverse primer (5'-3'): CAAATAGCCTGGAGAACTGCCTGAC
  * Normalization using housekeeping gene (GAPDH) Forward primer (5'-3'): GAAACCTGCCAAGTATGATG Reverse primer (5'-3'): AGGAAATGAGCTTGACAAAG 2-Assesment of CCL20 plasma level
  * Using Enzyme Linked Immunosorbent Assay kit (ELISA).

SUMMARY:
Rheumatoid arthritis (RA) is characterized as a systemic auto immune disorder linked to a persistent inflammatory process that can harm both joints and extra articular organs.

The upregulation of the CCR6/CCL20 axis in the synovial tissues and salivary glands (in cases of secondary Sjögren's syndrome) is considered to contribute to the recruitment of Th17 cells, which in turn enhances IL 17A production and promotes the inflammatory cycle.

DETAILED DESCRIPTION:
Although the aetiology and progression of RA remain incompletely elucidated, various therapeutic modalities are accessible, significantly altering the prognosis of patients with the disease.

Various cell types are implicated in the pathophysiology of RA, including synovial fibroblasts, osteoclasts, immune associated T and B lymphocytes, and macrophages. The orchestration of these cells induces the release of diverse inflammatory mediators (cytokines and chemokines) that perpetuate the chronic inflammatory response of the disease. Chemokines and their receptors regulate lymphocyte recruitment to inflamed joints in RA. Cytokines, encompassing both pro inflammatory and anti-inflammatory types, are recognized for their essential involvement in the evolution of RA via inflammation and the degradation of articular cartilage.

The chemokine receptor (CCR)6 is a class A GPCR within the chemokine family, noted for its notable therapeutic promise in immunological research.

The sole chemokine ligand for CCR6 is chemokine ligand 20 (CCL20), which is also referred to as macrophage inflammatory protein (MIP) 3α, Exodus 1 and liver and activation regulated chemokine. In humans, it is expressed by neutrophils, Th17 cells and peripheral blood mononuclear cells. This axis has distinct functions in immunological homeostasis and activation.

CCL20 is one of the chemokines mainly produced by inflamed synovial cells in response to cytokines, including TNF-α (tumour necrosis factor-α), IL-1, IL-17, and IL-18.

Synovial T lymphocytes generate cytokines, such as TNFα, IFNγ and IL 17A. The production of pro inflammatory cytokines was originally ascribed to Th1 cells Subsequently, it was elucidated that IL 17A production among Th cells was confined to a distinct Th cell subpopulation, subsequently designated as Th17.

The interaction between CCR6 and CCL20 is critical, not only for the migration of Th17 cells, but also for their activation and differentiation. CCL20 has been shown to be involved in the differentiation of naive T cells into Th17 cells, thereby directly influencing IL 17A production in patients with RA.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-60 years) diagnosed with RA according to the American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) 2010 classification criteria for RA by an expert rheumatologist.

Exclusion Criteria:

* • Patients with co-existing infections or other autoimmune diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with Rheumatoid Arthritis aged from 18 years to 60 years, in Rheumatology and Rehabilitation department of Sohag University Hospital and healthy controls of matched age and sex
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
assess expression of CCR6 gene in peripheral blood leukocytes of RA patients compared to healthy individuals | within 3 days of samples collection
  assessment of CCR6 gene expression level using quantitative real time PCR

SECONDARY OUTCOMES:
Measure the plasma levels of CCL20 | within 3 days after samples collection
  Measurement of the plasma levels of CCL20 using enzyme-linked immunosorbent assay (ELISA)

REFERENCES:
- [Background] Conforti A, Di Cola I, Pavlych V, Ruscitti P, Berardicurti O, Ursini F, Giacomelli R and Cipriani P (2021): Beyond the joints, the extra-articular manifestations in rheumatoid arthritis. Autoimmun Rev 20: 102735.
- [Background] 2- Ciofani M, Madar A, Galan C, Sellars M, Mace K, Pauli F, Agarwal A, Huang W, Parkhurst CN, Muratet M, et al (2012): A vali dated regulatory network for Th17 cell specification. Cell 151: 289-303.
- [Background] 1- Al Obaidi MJ and Al Ghurabi BH: Potential role of NLRP3 inflammasome activation in the pathogenesis of periodontitis patients with type 2 diabetes mellitus. J Med Chem Sci 6: 522-531, 2023.